CLINICAL TRIAL: NCT00571038
Title: Working With Veterans Organizations to Improve Blood Pressure
Acronym: POWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Medical College of Wisconsin (Other); Veterans of Foreign Wars USA (Other); Vietnam Veterans of America (Unknown); National Association of Black Veterans (Unknown); Korea Veterans of America, Inc. (Other); Disabled American Veterans (Other); AmVETS (Unknown); Jewish War Veterans of the United States of America (Other); The American Legion Department of Wisconsin (Other); Wisconsin Elks Association (a branch of The Benevolent and Protective order of Elks of the United States of America) (Unknown)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IAB 06-086
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
Keywords: Hypertension; Self-help groups; Community health networks; Health knowledge, attitudes, practice; Patient participation; Randomized clinical trial
MeSH Terms: conditions — Hypertension; Behavior; Patient Participation | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer Led (Experimental): Post provided with blood pressure cuffs, pedometers and scale. Two post members trained as peer leaders who encourage post members to take positive steps to improve BP. Peer leader training involves 20 hours of training over 12 months, telephone/email access to clinical experts and educational materials to share with post members.
  Interventions: Behavioral: Peer Led
- Seminar (Active Comparator): Post provided with blood pressure cuffs, pedometers and scale. Post members, including study participants invited to didactic sessions on cardiovascular health.
  Interventions: Behavioral: Seminar

INTERVENTIONS:
Behavioral: Peer Led — Post provided with blood pressure cuffs, pedometers and scale. Two post members trained as peer leaders who encourage post members to take positive steps to improve BP. Peer leader training involves 20 hours of training over 12 months, telephone/email access to clinical experts and educational materials to share with post members.
  Other Names: Peer led education and support
  Arms: Peer Led
Behavioral: Seminar — Post provided with blood pressure cuffs, pedometers and scale. Post members, including study participants invited to didactic sessions on cardiovascular health.
  Other Names: Professional didactic education
  Arms: Seminar

SUMMARY:
The primary purpose of this project is to establish the efficacy of a novel peer support intervention to reduce hypertension among members of veteran service organizations (VSOs). Specifically, we plan to demonstrate that veterans participating in a peer support intervention, as opposed to a purely didactic educational program, will have better blood pressure (BP) control, increased engagement in blood pressure lowering activities (such as exercise), and a more active stance as patients.

DETAILED DESCRIPTION:
IMPACT ON VETERANS HEALTH It is anticipated that this intervention will help participating veterans achieve optimal hypertension (HTN) control. Doing so will reduce their risks for heart disease and stroke, and improve their quality of life. It is hoped that the collaborative nature of this intervention will strengthen the Department of Veterans Affairs (VA)'s ties to the veteran community, and establish important "partnerships for health." If successful, this intervention could serve as a model for managing chronic disease both within and outside the VA system.

BACKGROUND/RATIONALE Despite consensus that effective hypertension treatment reduces morbidity and mortality, many patients in the United States continue to have suboptimal blood pressure control. Even with the provider resources and motivated patients inherent in a randomized clinical trial, over a third of patients participating in the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT) were not at their goal blood pressure of 140/90 after five years. Similarly, within the Veterans Integrated Service Network (VISN) 12 we have found that as many as 30% of patients with hypertension are above the target BP of 140/90, despite routine physician reminders to patients who are above these goals. Moreover, preliminary results of an internally funded randomized trial suggest minimal impact of further physician-focused interventions to reduce patients' blood pressure.

OBJECTIVES We will have two primary objectives. First, because the intervention proposed is novel, we believe we need to demonstrate its efficacy in a methodologically rigorous fashion. Specifically we plan to demonstrate that veterans participating in a peer support intervention will have improved blood pressure control, knowledge of blood pressure treatment, both generally and for themselves, and a more active stance as patients.

Second, we will carefully examine the process by which our intervention achieves these goals, including examining such key structural variables as the frequency of peer support meetings, attendance of participants at these meetings, and use of healthcare professional support by the group leaders. As part of this second objective, we also seek to understand the fidelity with which the peer leaders are to deliver the intervention, and the satisfaction of both support group participants and leaders with the intervention.

METHODS There are three primary activities in the present project.

First, academicians from the Clement J. Zablocki VA Medical Center (VAMC) are working with the Veterans of Foreign Wars (VFW) and other community groups to develop a community-academic partnership that follows the principles of community-based participatory research. This key activity is underway and will continue beyond the present period of funding. Second, the centerpiece of the present grant is a cluster randomized clinical trial (RCT) of the use of peer-led support groups to improve BP control in patients with hypertension. Fifty posts drawn from the VFW, American Legion, Vietnam Veterans Association, and National Association of Black Veterans will be randomly assigned to receive professionally delivered education regarding hypertension or to a peer support intervention. The third activity is an evaluation of the processes involved in delivering the peer support intervention that will allow for successful replication, or to provide insight into why the expected improvement in BP control did not occur.

ELIGIBILITY:
Inclusion Criteria:

1. Member of a post or auxiliary of a participating veterans' service organization or Elks Lodge in the 70 miles surrounding the Milwaukee VAMC.
2. Hypertension as established by one of: a) Average systolic blood pressure (SBP) greater than 140 or diastolic blood pressure (DBP) greater than 90 at two baseline visits; b) SBP greater than 130 or DBP greater than 90 at two baseline visits, plus patient report of diabetes mellitus and use of a hypoglycemic agent at the baseline visit; or c) self-reported hypertension plus self-reported current treatment with at least one antihypertensive drug at baseline visit.
3. Willingness to sign informed consent document.

Exclusion Criteria:

1. Medical or social condition preventing routine attendance at a monthly meeting.
2. Inability to communicate with other post members because of language barrier or physical limitation (e.g., prior stroke).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Whittle, MD MPH, Principal Investigator — Clement J. Zablocki VA Medical Center, Milwaukee, WI
Locations (1):
- Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Rosenwald K, Ertl K, Fletcher KE, Whittle J. Patterns of arthritis medication use in a community sample. J Prim Care Community Health. 2012 Oct 1;3(4):272-7. doi: 10.1177/2150131912442388. Epub 2012 Apr 4. PMID 23804172
- [Background] Patterson L, Morzinski J, Ertl K, Wurm C, Hayes A, Whittle J. Engaging community-based veterans' organizations in health promotion programs. Fam Community Health. 2011 Oct-Dec;34(4):311-8. doi: 10.1097/FCH.0b013e31822b5425. PMID 21881418
- [Background] Whittle J, Fletcher KE, Morzinski J, Ertl K, Patterson L, Jensen W, Schapira MM. Ethical challenges in a randomized controlled trial of peer education among veterans service organizations. J Empir Res Hum Res Ethics. 2010 Dec;5(4):43-51. doi: 10.1525/jer.2010.5.4.43. PMID 21133786
- [Background] Shirk J, Fletcher K, Patterson L, Grippen A, Eastwood D, Whittle JC. Peer leader characteristics do not predict their ability to deliver a peer support intervention. [Abstract]. Journal of general internal medicine. 2010 Jul 1; 25(Supple 3):S347.
- [Background] Hayes A, Morzinski J, Ertl K, Wurm C, Patterson L, Wilke N, Whittle J. Preliminary description of the feasibility of using peer leaders to encourage hypertension self-management. WMJ. 2010 Apr;109(2):85-90. PMID 20443327
- [Result] Whittle J, Schapira MM, Fletcher KE, Hayes A, Morzinski J, Laud P, Eastwood D, Ertl K, Patterson L, Mosack KE. A randomized trial of peer-delivered self-management support for hypertension. Am J Hypertens. 2014 Nov;27(11):1416-23. doi: 10.1093/ajh/hpu058. Epub 2014 Apr 22. PMID 24755206
- [Result] Whittle JC, Hayes A, Eastwood D, Morzinski J, Ertl K, Wurm C. Effect on health behaviors of a health promotion intervention delivered through veterans service organizations. [Abstract]. Journal of general internal medicine. 2010 Jul 1; 25(Supple 3):S264.
- See also: Click here for more information about this study: Working with Veterans Organizations to Improve Blood Pressure — http://www.milwaukee.va.gov/Power/Power.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We wrote letters to posts located within 60 miles of the study hospital and followed up with a phone call to arrange for an in-person presentation. Before and after the presentation, we measured blood pressures and asked about diagnoses of hypertension. We scheduled individual appointments with potential subjects to confirm eligibility and consent.
Pre-assignment Details: Posts had to identify two potential peer leaders to be eligible for the trial. The post membership voted on whether to participate, even though many would not be followed as study members. All enrollment activities occurred before posts were assigned to an intervention. All participants within a post received the assigned intervention.
Groups:
- Seminar: Post provided with blood pressure cuffs, pedometers and scale. Post members, including study participants invited to didactic sessions on cardiovascular health. Two or more post representatives (who were also post members) coordinated use of equipment and encouraged members to attend the didactic sessions.
Period: Overall Study
Arm/Group | Peer Led | Seminar
Started | 219 | 185
6 Month Follow up | 208 | 176
18 Month Survey Only | 199 | 163
Completed | 208 (7 died 2 moved 1 asked to be withdrawn 1 unable to reach) | 171 (5 died 2 moved 3 asked to be withdrawn 4 unable to reach)
Not Completed | 11 | 14
Not completed — Lost to Follow-up | 1 | 4
Not completed — Death | 7 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Moved out of state | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Led | Seminar | Total
Number analyzed (Participants) | 219 | 185 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (9.97) | 67.4 (10.3) | 68.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 17 | 51
  Male | 185 | 168 | 353
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 8 | 11
  White | 214 | 175 | 389
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 219 | 185 | 404

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure
Description: Mean/Standard Error (SE) change in systolic blood pressure
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 208 | 171
mm Hg | -3.48 (1.13) | -5.45 (1.24)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.2417, Mixed Models Analysis

2. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Mean/SE change in diastolic blood pressure
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 208 | 171
mm Hg | -1.83 (0.76) | -2.03 (0.83)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.8586, Mixed Models Analysis

3. Secondary Outcome: Change in Weight
Description: Mean/SE change in weight, measured in pounds (lbs)
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: pounds
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 208 | 171
pounds | -0.85 (0.71) | 1.29 (0.78)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.0432, Mixed Models Analysis

4. Secondary Outcome: Change in BMI
Description: Mean/SE change in Body Mass Index (BMI) (kg/m2)
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 208 | 171
kg/m2 | -0.12 (0.10) | 0.17 (0.12)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.0604, Mixed Models Analysis

5. Secondary Outcome: Change in Health Status
Description: Response to the question "How would you rate your general health status?". Response options are scored as follows.
  1. Excellent
  2. Very Good
  3. Good
  4. Fair
  5. Poor We report the change in health status from baseline to 12 months.
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: units on a scale (range 1-5)
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
units on a scale (range 1-5) | -0.14 (0.052) | 0.018 (0.054)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.0438, Kruskal-Wallis

6. Secondary Outcome: Change in Time Since Last Physician Visit
Description: Change in mean # of months since last visit to a physician
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: months (since last visit)
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
months (since last visit) | -2.58 (0.409) | -1.65 (1.049)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.1418, Kruskal-Wallis

7. Secondary Outcome: Non-Clinic Blood Pressure Checks
Description: % reporting non-clinic blood pressure (BP) checks at least once a month
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Number; unit: percentage of participants
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
percentage of participants | 91.26 | 82.74
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.0070, Fisher Exact; Two-sided Pr <= P

8. Secondary Outcome: Change in Number of Blood Pressure Medications
Description: Change in mean # of prescription blood pressure medications
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: blood pressure medications
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
blood pressure medications | 0.011 (0.054) | 0.028 (0.057)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.8395, Kruskal-Wallis

9. Secondary Outcome: Change in Hypertension Knowledge
Description: Mean/SE change in score on:
  Scale: Hypertension Evaluation of Lifestyle and Management (HELM) Construct: Knowledge of hypertension and lifestyle factors related to hypertension Minimum Score: 0 Maximum Score: 14 Interpretation of Score: Higher is better
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | 0.529 (0.127) | 0.256 (0.159)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.2194, Kruskal-Wallis

10. Secondary Outcome: Change in Hypertension Attitudes
Description: Mean/SE change in score on:
  Scale: Not applicable; series of agree/disagree statements that we wrote Construct: Attitudes around blood pressure diagnosis, treatment (including lifestyle changes), and seriousness of the condition Minimum Score: 12 Maximum Score: 60 Interpretation of Score: Lower is better
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | -0.24 (0.292) | -0.19 (0.307)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.9191, Kruskal-Wallis

11. Secondary Outcome: Change in Satisfaction With Blood Pressure Treatment
Description: Mean/SE change in score on:
  Scale: Modified Holmes-Ravnor Satisfaction with Decision (SWD) Construct: Satisfaction with current blood pressure treatment Minimum Score: 1 Maximum Score: 5 Interpretation of Score: Lower is better (NOTE: Original instrument's scoring is reversed; i.e., higher is better)
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | -0.15 (0.052) | -0.15 (0.058)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.9633, Kruskal-Wallis

12. Secondary Outcome: Change in Alcohol Use
Description: Mean/SE change in score on:
  Scale: Alcohol Use Disorders Identification Test (AUDIT) Construct: Alcohol use and abuse Minimum Score: 0 Maximum Score: 12 Interpretation of Score: Lower is better
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | -0.15 (0.097) | -0.19 (0.128)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.5901, Kruskal-Wallis

13. Secondary Outcome: Change in Sodium Intake
Description: Mean/SE change in score on:
  Scale: Hopkins Dietary Questionnaire (only the dietary salt avoidance questions) Construct: Dietary sodium intake Minimum Score: 2 Maximum Score: 12 Interpretation of Score: Higher is better
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | -0.08 (0.159) | -0.11 (0.166)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.9820, Kruskal-Wallis

14. Secondary Outcome: Change in Physical Activity Level
Description: Mean/SE change in score on:
  Scale: International Physical Activity Questionnaire (IPAQ), Metabolic Equivalent of Task (MET) Construct: Total metabolic equivalents (a measure of energy expenditure) in the last 7 days Minimum Score: 0 Maximum Score: Not applicable; based on physical activity done Interpretation of Score: Higher is better
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: METS
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
METS | 260.2 (321.9) | -89.5 (409.3)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.3979, Kruskal-Wallis

15. Secondary Outcome: Change in Daily Steps
Description: Mean/SE change in # of steps per day (self report)
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: steps per day
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
steps per day | 2395 (875.5) | 963.5 (735.9)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.1471, Kruskal-Wallis

16. Secondary Outcome: Change in Fruit and Vegetable Intake
Description: Mean/SE change in # of servings per day; questions taken from the 2009 Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: servings of fruits & vegetables per day
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
servings of fruits & vegetables per day | 0.096 (0.109) | -0.01 (0.093)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.6123, Kruskal-Wallis

17. Secondary Outcome: Change in Medication Adherence
Description: Mean/SE change in score on:
  Scale: Morisky Adherence; questions modified to ask specifically about blood pressure medication Construct: Adherence to prescribed medication-taking regimen Minimum Score: 0 Maximum Score: 4 Interpretation of Score: Lower is better
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | -0.02 (0.043) | 0.007 (0.055)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.5861, Kruskal-Wallis

18. Secondary Outcome: Change in Self Efficacy
Description: Mean/SE change in score on:
  Scale: Schwarzer General Perceived Self-Efficacy Construct: Perceived self-efficacy Minimum Score: 10 Maximum Score: 40 Interpretation of Score: Higher is better
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | 0.450 (0.246) | 0.286 (0.275)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.4489, Kruskal-Wallis

19. Secondary Outcome: Change in Social Support
Description: Mean/SE change in overall score on:
  Scale: Medical Outcomes Study (MOS) Social Support Survey Construct: Overall measure of social support, including tangible, affectionate, positive social interaction, and emotional/informational Minimum Score: 0 Maximum Score: 100 Interpretation of Score: Higher is better
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | 1.249 (1.088) | 2.227 (1.171)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.2527, Kruskal-Wallis

20. Secondary Outcome: Change in Health Opinions
Description: Mean/SE change in overall score on:
  Scale: Krantz Health Opinion Survey Construct: Opinions about healthcare and healthcare providers Minimum Score: 0 Maximum Score: 16 Interpretation of Score: Higher is better
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | 0.252 (0.167) | 0.232 (0.188)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.7314, Kruskal-Wallis

21. Secondary Outcome: Change in Patient Activation
Description: Mean/SE change in score on:
  Scale: Hibbard Patient Activation Measure (PAM) Construct: Level of patient activation and engagement in health care Minimum Score: 0 Maximum Score: 100 Interpretation of Score: Lower is better (NOTE: Original instrument's scoring is reversed; i.e., higher is better)
Time Frame: 9/16/2008-8/9/2010; baseline and 12 months
Population: Consented, hypertensive members of participating veterans service organizations in SE Wisconsin.
Measure: Mean (Standard Error); unit: survey score
Arm/Group | Peer Led | Seminar
Number analyzed (Participants) | 206 | 168
survey score | 1.007 (0.903) | 1.254 (0.910)
Statistical Analysis 1: Comparison: Peer Led vs Seminar; Test type: Superiority or Other; p = 0.9839, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 2 years (2009-2011)
Arm/Group | Peer Led | Seminar
Serious Adverse Events (participants affected / at risk) | 17/219 | 8/185
Other Adverse Events (participants affected / at risk) | 0/219 | 0/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Led (N=219) | Seminar (N=185)
Death (General disorders) | 9 (9) | 5 (5)
Hospitalization (General disorders) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 3 (3) | 1 (1)
Stroke (Vascular disorders) | 1 (1) | 2 (2)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Cancer (General disorders) | 1 (1) | 0 (0)
ER Visit (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes